CLINICAL TRIAL: NCT03975452
Title: Phase II Study on Volume De-escalation in Neoadjuvant Radiochemotherapy of Rectal Cancer
Brief Title: Volume De-escalation in Neoadjuvant Radiochemotherapy of Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Michele Fiore, MD, Researcher, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8/07 PAR ComEt CBM
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Toxicity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary resectable cT2-low lying-T3, N0-N1 rectal tumour (Experimental): Primary resectable cT2-low lying-T3, N0-N1 adenocarcinoma of the rectum, without evidence of disease in lateral lymph nodes.
  Interventions: Radiation: Reduced radiation volumes

INTERVENTIONS:
Radiation: Reduced radiation volumes — Patient treated with reduced radiation volumes with the exclusion of elective pelvic nodal irradiation

SUMMARY:
The study outlines a clinical prospective protocol consisting of preoperative chemoradiation in locally advanced rectal cancer, without elective pelvic nodal irradiation. The proposal to exclude lateral spaces from the target volume is based on the assumption that the radiological evidence of recurrence in the lateral lymph nodes is shown to be below 5%. In the study all patients underwent an accurate pre-treatment work-up including total body CT, pelvic MRI and 18-fluorodeoxyglucose PET/CT, in order to include patients without evidence of disease in lateral lymph nodes. The primary endpoint of the study was the reduction of gastrointestinal toxicity; secondary endpoints were the pathological complete response (pCR), the local control (LC) rate, the overall survival (OS) and the disease-free survival (DFS).

DETAILED DESCRIPTION:
Patients affected by histologically proven rectal cancer were considered for enrollment in a prospective protocol that included preoperative CRT and surgical treatment. All patients underwent pre-treatment work-up (clinical examination, pancolonoscopy with biopsy, total body CT scan, pelvic MRI, and whole body 18-fluorodeoxyglucose PET/CT scan). Eligible patients had primary resectable cT2-low lying-T3, N0-N1 adenocarcinoma of the rectum, without evidence of disease in lateral lymph nodes. Additional eligibility criteria included performance status as well as liver, kidney, and bone marrow function that allowed for long-course CRT, older than 18 years, and no distant metastases.

ELIGIBILITY:
Inclusion Criteria:

* Primary resectable cT2-low lying-T3, N0-N1 adenocarcinoma of the rectum, without evidence of disease in lateral lymph nodes
* No distant metastases

Exclusion Criteria:

* Evidence of disease in lateral lymph nodes
* Distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The reduction of gastrointestinal (GI) toxicity | 36 months
  The study is planned to obtain a 66% reduction in acute grade 3 or higher GI side-effects

SECONDARY OUTCOMES:
Pathological complete response (pCR) | 36 months
  All study sample characteristics will be summarized with descriptive statistics
The local control (LC) rate | 36 months
  The LC will be calculated by the Kaplan-Meier method. Evaluation of differences will be performed with the log-rank test. Survival will be censored at the time of the last follow-up or death. A two-sided P value of 0.05 will be considered significant.
The overall survival (OS) | 36 months
  The OS will be calculated by the Kaplan-Meier method. Evaluation of differences will be performed with the log-rank test. Survival will be censored at the time of the last follow-up or death. A two-sided P value of 0.05 will be considered significant.
The disease-free survival (DFS) | 36 months
  The DFS will be calculated by the Kaplan-Meier method. Evaluation of differences will be performed with the log-rank test. Survival will be censored at the time of the last follow-up or death. A two-sided P value of 0.05 will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Trodella, Prof, Principal Investigator — Campus Bio-Medico University
Locations (1):
- Michele Fiore, Rome, Italy

IPD SHARING:
Plan to Share IPD: No